CLINICAL TRIAL: NCT00124111
Title: A Single-arm Study Evaluating the Relative Dose Intensity of IV CMF Given on Day 1 and Day 8 With Pegfilgrastim Support in Subjects With Stage I-III Breast Cancer
Brief Title: A Study of Cyclophosphamide/Methotrexate/5-Fluorouracil (CMF) With Pegfilgrastim in Subjects With Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Global Development Leader, Amgen Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: 20030156
Record Dates: First submitted 2005-07-25; First posted 2005-07-27 (Estimated); Last update posted 2010-02-26 (Estimated); Status verified 2010-02

CONDITIONS: Breast Cancer
Keywords: clinical trial; pegfilgrastim; haematopoietic growth factor; neutropenia; CMF; Cancer
MeSH Terms: conditions — Breast Neoplasms; Neutropenia; Neoplasms | interventions — pegfilgrastim; Cyclophosphamide; Methotrexate; Fluorouracil

INTERVENTIONS:
Drug: pegfilgrastim
Drug: cyclophosphamide
Drug: methotrexate
Drug: 5-fluorouracil

SUMMARY:
The purpose of this study is to assess the relative dose intensity (RDI) of intravenous (IV) CMF on a Day 1 and 8 schedule given every 28 days with pegfilgrastim support in subjects with stage I-III breast cancer.

ELIGIBILITY:
Inclusion Criteria: - Histologically confirmed breast cancer Stage I, II or III - Candidate for IV CMF chemotherapy (every 4 weeks) for a total of 6 cycles - Chemotherapy naïve (prior treatment with hormone therapy or with anti-HER2 monoclonal antibody therapy is permitted as long as treatment has been stopped prior to enrollment into the study) - Absolute neutrophil count (ANC) greater than or equal to 1.5 x 10^9/L - Platelet count greater than or equal to 100 x 10^9/L - Eastern Cooperative Oncology Group (ECOG) performance status of 0-2 - Written informed consent before any study specific procedure Exclusion Criteria: - AST and/or ALT greater than 1.5 x upper limit of normal (ULN) concomitant with alkaline phosphatase greater than 2.5 x ULN according to institutional standard - Bilirubin greater than 2 x ULN according to institutional standard - Inadequate renal function (creatinine greater than 1.5 x ULN according to institutional standard) - Any premalignant myeloid condition or any malignancy with myeloid characteristics (e.g., myelodysplastic syndromes, acute or chronic myelogenous leukaemias) - History of prior malignancy other than breast cancer with the exception of curatively treated basal cell or squamous cell carcinoma of the skin, in situ cervical carcinoma, or other surgically cured malignancy - Prior radiotherapy - Scheduled concomitant radiotherapy (e.g., radiotherapy administration while on study) - Documented active infection at the time of enrolment requiring use of systemic anti- infectives - Documented positive test for human immunodeficiency virus (HIV) infection - Known hypersensitivity to E coli derived products [e.g., Filgrastim (Neupogen®), pegfilgrastim (Neulasta®), HUMULIN® Insulin, L-Asparaginase, HUMATROPE® Growth Hormone, INTRON A®] - Subject is currently enrolled in or 30 days have not passed since completing other investigational device or drug trial(s) or is receiving other investigational agent(s) other than placebo (confirmation of prior treatment must be documented) - Pregnant or breast-feeding (for subjects of child bearing potential) - Not using adequate contraception (for subjects of child bearing potential) - Previous participation in this study - Inability or unwillingness to comply with the protocol procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

PRIMARY OUTCOMES:
To assess the relative dose intensity (RDI) of IV CMF Day 1 and 8 schedule given every 28 days with pegfilgrastim support in subjects with Stage I-III breast cancer.

SECONDARY OUTCOMES:
Incidence of febrile neutropenic events over all cycles
Incidence of dose delays and dose reductions of planned chemotherapy due to neutropenic events
Safety profile over all cycles

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Result] Mattioli R, Gridelli C, Castellanos J, Duque A, Falcone A, Mansutti M, Bacon P, Lawrinson S, Skacel T, Casas A. Use of pegfilgrastim support on day 9 to maintain relative dose intensity of chemotherapy in breast cancer patients receiving a day 1 and 8 CMF regimen. Clin Transl Oncol. 2009 Dec;11(12):842-8. doi: 10.1007/s12094-009-0453-4. PMID 20045791
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com
- See also: Notice regarding posted summaries of trial results — http://download.veritasmedicine.com/REGFILES/amgen/Amgen_results_disclaimer.pdf
- See also: To access clinical trial results information click on this link — http://download.veritasmedicine.com/REGFILES/amgen/08D_FDAMA_113_Posting_Summary_11_GCSFSD01_20030156.pdf
- See also: FDA-approved Drug Labeling — http://www.neulasta.com/